CLINICAL TRIAL: NCT02831270
Title: Does Acute Normovolemic Hemodilution Affect Intraoperative Value of Serum-creatinine Concentration in Patients Undergoing Cardiac Surgery?
Brief Title: Acute Normovolemic Hemodilution on Serum-creatinine Concentration in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Other Study IDs: KUH1160004-1
Record Dates: First submitted 2016-07-10; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Mitral Regurgitation; Mitral Stenosis; Tricuspid Regurgitation
Keywords: cardiac surgery; acute normovolemic hemodilution
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis; Tricuspid Valve Insufficiency | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: Patients undergoing cardiac surgery supposed not to get acute normovolemic hemodilution (ANH) before CPB
- Active Comparator: Acute normovolemic hemodilution group: Patients undergoing cardiac surgery supposed to get aucte normovolemic hemodilution (ANH) before CPB
  Interventions: Procedure: Acute normovolemic hemodilution (ANH); Drug: hydroxyethyl starch (HES 130/0.6)

INTERVENTIONS:
Procedure: Acute normovolemic hemodilution (ANH)
  Groups: Active Comparator: Acute normovolemic hemodilution group
Drug: hydroxyethyl starch (HES 130/0.6)
  Groups: Active Comparator: Acute normovolemic hemodilution group

SUMMARY:
Serum-creatinine level (s-Cr) is an important factor for predicting perioperative patient's outcome regarding acute kidney injury. Although cardiopulmonary bypass (CPB), an essential procedure for cardiac surgery, dilutes patient's blood components, possible impact of applying acute normovolemic hemodilution (ANH) and CPB on s-Cr has not been well investigated.

In patients undergoing cardiac surgery employing moderate hypothermic CPB (age 20-71 years, n=32), ANH will be randomly applied to 15 patients (Group-ANH) but not in 17 patients (Group-C) before initiating CPB. For ANH procedure consisting of 5 ml/kg of blood salvage and administering 5 ml/kg of balanced hydroxyethyl starch (HES) 130/0.4 for 15 min will be started at 30 min after anesthesia induction and before CPB application for surgery. In both groups, moderate hypothermic CPB will be initiated by using 1600-1800 ml of bloodless priming solution. The changes of hematocrit (Hct), Na+, K+, HCO3-, Ca2+, osmolarity, s-Cr will be determined before ANH (T1), after the first ANH of 2.5 ml/kg (T2), and after the second ANH of 2.5 ml/kg (T3), 30 sec and 60 sec after the initiation of CPB (T4, T5), immediately and 1 hour after the weaning from CPB (T6, T7) and at the end of surgery (T8). S-Cr will be determined by using a point-of-care test device (StatSensor™ Creatinine, Nova Biomedical, USA).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery with cardiopulmonary bypass who signed written informed consent

Exclusion Criteria:

* preoperative renal failure requiring reran replacement therapy
* preoperative liver disease
* preoperative low cardiac output (EF < 50%)
* Preoperative IABP application, Atrial fibrillation, Pacemaker,
* contraindication for applying TEE
* intraoperative withdrawal

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery due to valvular heart disease
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
serum creatinine (s-Cr) concentration | before ANH

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea